CLINICAL TRIAL: NCT06725641
Title: Bioequivalence Study of Methacholine for Inhalation
Brief Title: Bioequivalence Study of Methacholine for Inhalation (pharmacodynamics)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ting YANG, Principal Investigator, China-Japan Friendship Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: TQC3610-BE-01(PD)
Record Dates: First submitted 2024-11-30; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Asthma
Keywords: Clinically diagnosed asthma patients or other individuals willing to undergo bronchial provocation tests.
MeSH Terms: conditions — Asthma | interventions — Inhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test preparation：Methylcholine chloroacetate for inhalation (Experimental): Inhale different concentrations of choline chloride solution
  Interventions: Drug: Test preparation：Methylcholine chloroacetate for inhalation
- Reference preparation：Methylcholine chloroacetate for inhalation（Provocholine） (Active Comparator): Inhale different concentrations of choline chloride solution
  Interventions: Drug: Reference preparation：Methylcholine chloroacetate for inhalation（Provocholine）

INTERVENTIONS:
Drug: Test preparation：Methylcholine chloroacetate for inhalation — Cholinergic agonists
  Arms: Test preparation：Methylcholine chloroacetate for inhalation
Drug: Reference preparation：Methylcholine chloroacetate for inhalation（Provocholine） — Cholinergic agonists
  Arms: Reference preparation：Methylcholine chloroacetate for inhalation（Provocholine）

SUMMARY:
This trial was divided into two parts. This is the scecond part. The second part is the pharmacodynamic equivalence study of patients, which is a single-dose, randomized, open, two-cycle, two-sequence crossover design, and plans to enroll 40 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. adults 18 years old ≤ age ≤65 years old, gender is not limited.
2. Lung function test FEV1≥70% of the predicted value, and FEV1/FVC≥0.7. 3. Patients with clinically diagnosed asthma or others willing to accept bronchial stimulation test.

4. Patients who use contraindicated drugs (β2 adrenergic receptor agonists, anticholinergics, oral bronchodilators, antihistamines, leukotriene receptor antagonists) may be discontinued during the prescribed period prior to airway reactivity examination.

5, voluntary enrollment, signed informed consent, compliance is good, can cooperate with the test observation.

Exclusion Criteria:

1. there is a history of allergy to this reagent.
2. Patients with a history of heart disease who have difficulty tolerating bronchial provocation tests.
3. Patients who had received thoracic or abdominal surgery within 6 months before the trial.
4. Patients who had undergone surgery for intracranial, eye, ear, nose and throat, and respiratory diseases within 6 months before the trial.
5. Patients with respiratory diseases such as pneumothorax or infectious diseases such as tuberculosis.
6. Patients with diseases that may be affected by the use of cholinergic drugs (epilepsy, bradycardia, coronary artery occlusion, vagus nerve tension, thyroid disease, arrhythmia, peptic ulcer, urinary tract disorders, etc.).
7. Patients with a history of drug dependence or alcohol dependence.
8. Severe circulatory system diseases, liver and bile system diseases, digestive tract diseases, urinary system diseases, kidney diseases, blood diseases, endocrine system diseases, immune system diseases, malignant tumors, etc.
9. Patients who are taking cholinase inhibitors (for myasthenia gravis).
10. Patients with unexplained urticaria.
11. Pregnant and lactating women.
12. The subjects had dyspnea, wheezing or wheezing on the test day.
13. have myocardial infarction or stroke, combined with hypertension (systolic blood pressure >200mmHg, diastolic blood pressure >100mmHg) patients.
14. Poor coordination of basic lung function examination and failure to meet quality control.
15. Patients who have used drugs that affect airway contractile function and airway inflammation before the trial and can not be stopped (bronchodilators, glucocorticoids, antiallergens and triene receptor antagonists, etc.).
16. Current smokers, those who had quit smoking for less than one year at the time of screening, and those who had a smoking history of more than 10 pack-years.
17. Patients admitted to hospital for exacerbation of asthma within 12 weeks.
18. combined with patients with respiratory diseases (such as COPD) that may affect the efficacy and safety evaluation of the drug.
19. Researchers believe that there are any cases that are not suitable for inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-24 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-26 (Actual)

PRIMARY OUTCOMES:
Cumulative dose of inhaled activator with a 20% reduction in forced expiratory volume in the first second from baseline | 30 to 90 seconds after administration
  Cumulative dose of inhaled activator with a 20% reduction in forced expiratory volume in the first second from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ting Yang, Doctor, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-japan Friendship Hospital, Beijing, Beijing Municipality, China